CLINICAL TRIAL: NCT04580134
Title: Antipsychotic Response to Clozapine in B-SNIP Biotype-1 (Clozapine)
Brief Title: CLOZAPINE Response in Biotype-1
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Beth Israel Deaconess Medical Center (Other); Hartford Hospital (Other); University of Georgia (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Carol A. Tamminga, Chair, Department of Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ( STU-2020-0989 )
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar 1 Disorder
Keywords: Schizophrenia, Bipolar, Psychosis, Biomarker, Biotype, BSNIP, B-SNIP, IEA
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clozapine; Risperidone

STUDY DESIGN:
Intervention Model Description: Individuals who previously participated in a B-SNIP trial who have already been biotyped will be grouped accordingly.
  New incoming individuals will have their Biotype completed. Those with Biotypes 1 and 2 will be recruited into this protocol. Anyone with Biotype 3 will be excluded from this protocol, but their information will be retained for use in a later study.
  Biotypes 1 and 2 will be separated into two groups. Each Biotype, B1 and B2, will be randomized between risperidone and clozapine to create parallel comparator groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and those who interact with them are blinded to study medication. The pharmacy dispensing team and the Safety Officer will remain unblinded for safety reasons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Biotype 1 - Clozapine (B1C) (Experimental): Target doses will be up to clozapine 500mg po qd. In addition, several concomitant (open label) medications for symptomatic management will be available via the study protocol [non-benzodiazepine sleep aid (melatonin, hydroxyzine); motor side effect treatments (benztropine, propranolol)]. The doses for these medications will be consistent with those routinely used in a clinical practice: melatonin [up to 10mg at bedtime], hydroxyzine [up to 100mg at bedtime]; benztropine [up to 4mg/day (2mg twice/day)], propranolol [up to 40mg/day (20mg twice/day)].
  Interventions: Drug: clozapine
- Biotype 1 - Risperidone (B1R) (Placebo Comparator): Target doses will be up to risperidone 6mg po qd. In addition, several concomitant (open label) medications for symptomatic management will be available via the study protocol [non-benzodiazepine sleep aid (melatonin, hydroxyzine); motor side effect treatments (benztropine, propranolol)]. The doses for these medications will be consistent with those routinely used in a clinical practice: melatonin [up to 10mg at bedtime], hydroxyzine [up to 100mg at bedtime]; benztropine [up to 4mg/day (2mg twice/day)], propranolol [up to 40mg/day (20mg twice/day)].
  Interventions: Drug: risperidone
- Biotype 2 - Clozapine (B2C) (Active Comparator): Target doses will be up to clozapine 500mg po qd. In addition, several concomitant (open label) medications for symptomatic management will be available via the study protocol [non-benzodiazepine sleep aid (melatonin, hydroxyzine); motor side effect treatments (benztropine, propranolol)]. The doses for these medications will be consistent with those routinely used in a clinical practice: melatonin [up to 10mg at bedtime], hydroxyzine [up to 100mg at bedtime]; benztropine [up to 4mg/day (2mg twice/day)], propranolol [up to 40mg/day (20mg twice/day)].
  Interventions: Drug: clozapine
- Biotype 2 - Risperidone (B2R) (Placebo Comparator): Target doses will be up to risperidone 6mg po qd. In addition, several concomitant (open label) medications for symptomatic management will be available via the study protocol [non-benzodiazepine sleep aid (melatonin, hydroxyzine); motor side effect treatments (benztropine, propranolol)]. The doses for these medications will be consistent with those routinely used in a clinical practice: melatonin [up to 10mg at bedtime], hydroxyzine [up to 100mg at bedtime]; benztropine [up to 4mg/day (2mg twice/day)], propranolol [up to 40mg/day (20mg twice/day
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: clozapine — Biotype 1 and Biotype 2
  Other Names: Clozaril
  Arms: Biotype 1 - Clozapine (B1C); Biotype 2 - Clozapine (B2C)
Drug: risperidone — Biotype 1 and Biotype 2
  Other Names: Risperdal
  Arms: Biotype 1 - Risperidone (B1R); Biotype 2 - Risperidone (B2R)

SUMMARY:
The CLOZAPINE study is designed as a multisite study across 5 sites and is a clinical trial, involving human participants who are prospectively assigned to an intervention. The study will utilize a stringent randomized, double-blinded, parallel group clinical trial design. B2 group will serve as psychosis control with risperidone as medication control. The study is designed to evaluate effect of clozapine on the B1 participants, and the effect that will be evaluated is a biomedical outcome. The study sample will be comprised of individuals with psychosis, including 1) schizophrenia, 2) schizoaffective disorder and 3) psychotic bipolar I disorder. The investigators plan to initially screen and recruit n=524 (from both the existing B-SNIP library and newly-identified psychosis cases, ~50% each) in order to enroll n=320 (B1 and B2) into the RCT.

DETAILED DESCRIPTION:
The clinical hypotheses underlying this experiment are that (i) B1 individuals are uniquely responsive to the pharmacological properties of clozapine because they have low Intrinsic EEG Activity (IEA), an index of compromised cortical neuronal responsiveness. This is plausibly associated with both (ii) reduced excitatory and (iii) reduced inhibitory stimulation in cortex and that IEA will track this altered excitatory/inhibitory balance and parallel clinical antipsychotic response. Furthermore, (iv) B2 probands (based on their high IEA) will not respond to clozapine. In this study clozapine response is measured by a 'super-APD' (AntiPsychotic Drug) drug response, a response in addition to what is seen with a usual APD (e.g., risperidone). The investigators believe that the 30-35% of individuals who show a 'super-APD' clozapine response in schizophrenia in the pivotal study will be predominantly in B1, because the B1 completers will no longer be diluted by the other non-responders like B2s. Therefore, the investigators postulate that >50% of B1 will show a unique therapeutic action of clozapine (beyond general APD action), contrasted with the usual predicted response of B1 to risperidone or of B2 to clozapine or risperidone.

ELIGIBILITY:
Inclusion Criteria:

* 18-60y/o; males and females; all races and ethnicities; able to provide written informed consent; able to read, speak, and understand English; medically stable; meeting DSM-IV (SCID-based) criteria for schizophrenia, schizoaffective disorder, or bipolar I disorder with psychotic features (we will use DSM-IV to be consistent with prior B-SNIP samples); PANSS total score of ≥70 and at least one item scored ≥5 or two items scored ≥4 on PANSS Positive Subscale; normal baseline values for absolute neutrophil count (ANC above 1500/mm3)

Exclusion Criteria:

* premorbid intellectual ability estimate below 70 (WRAT-4, Word Reading subtest, age-corrected standardized score); comorbid DSM-IV diagnosis of alcohol or substance abuse in prior 1 month or substance dependence in prior 3 months; neurological (e.g., seizure disorder, stroke, traumatic brain injury with a loss of consciousness ≥ 30min) or severe medical condition (e.g., decompensated cardiovascular disorder, AIDS) that may affect central nervous system function; concomitant medications known to affect EEG properties (i.e., lithium, anticonvulsants, benzodiazepines) or strong CYP 1A2 inhibitors (e.g., ciprofloxacin, enoxacin) or strong CYP 3A4 inducers (e.g., phenytoin, carbamazepine, phenobarbital, rifampin) which cannot be safely discontinued; vulnerable populations (e.g., pregnant, nursing, incarcerated); unwilling to use reliable means of contraception; history of neuroleptic malignant syndrome; prior treatment with clozapine, prior treatment with long-acting injectable antipsychotics that are 1-month formulations within the past 3 months and for 3-month formulations within the past 6 months; intolerable side effects to either clozapine or risperidone in lifetime, or a previously failed trial of either clozapine or risperidone at adequate doses in lifetime; history of drug reaction with eosinophilia and systemic symptoms syndrome (DRESS), also known as drug-induced hypersensitivity syndrome (DIHS); high risk for suicide defined as more than 1 attempt in past 12 months that required medical attention, any attempt in the past 3 months or current suicidal ideation with plan and intent such that outpatient care is precluded; current homicidal ideation with plan and intent such that outpatient care is precluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 524 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in the PANSS total score | Week 4, Week 10 and Week 18
  The change in the PANSS total score from the clinical trial baseline (W4) to the end of treatment (W18) will be a primary outcome measure. We predict that B1/clozapine will show a significantly larger change in the PANSS score from W4 to W18, compared to B1/risperidone, B2/clozapine and B2/risperidone. We will also examine the patterns of change in the PANSS score during the 'stable treatment' phase (W10-W18), across the same study groups. A mixed-effect repeated-measures ANCOVA [2(Biotypes) × 2(clozapine/risperidone) × 2(time points] will be used. We also predict that the reduction in the PANSS scores will correlate with increased IEA in B1/clozapine but not in B1/risperidone, B2/clozapine or B2/risperidone. Multivariate prediction models will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Tamminga, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (5):
- United States (5):
  - Hartford Healthcare, Hartford, Connecticut
  - University of Georgia, Athens, Georgia
  - University of Chicago, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No